CLINICAL TRIAL: NCT06320977
Title: The Influence of Acute Static Stretching on the Ankle Joint-position Sense of Soccer Players: a Randomized Controlled Trial
Brief Title: The Influence of Acute Static Stretching on the Ankle Joint-position Sense of Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Fernando Pessoa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: ESS/FSA-397/23-2
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: Static Stretching; Joint Position Sense; Proprioception; Ankle; Soccer
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Condition (No Intervention): 5-minute rest
- Static Stretching of 30 seconds Condition (Active Comparator): Static stretching of the gastrocnemius and tibialis anterior muscles for 30 seconds
  Interventions: Other: Static Stretching
- Static Stretching of 90 seconds Condition (Active Comparator): Static stretching of the gastrocnemius and tibialis anterior muscles for 90 seconds
  Interventions: Other: Static Stretching

INTERVENTIONS:
Other: Static Stretching — The static stretching protocol will include the following muscle groups of the dominant lower limb:
  * Gastrocnemius - Participants will assume a bipedal position facing a wall. Then, the leg that is not being stretched will be placed forward, with the knee in semi-flexion, and the leg that is being stretched, behind, with the knee in full extension. Instructions will be given in order to keep the calcaneus on the floor;
  * Tibialis anterior - Participants will be facing a wall, with the entire foot in touch with the ground and toes pointing forward. Then, they will secure themselves to a handrail and project the hips back.
  These stretchings will be held in a position where the participants refer discomfort, and will be maintained for 30 seconds or 90 seconds according to the condition.
  Arms: Static Stretching of 30 seconds Condition; Static Stretching of 90 seconds Condition

SUMMARY:
The aim of this study isto investigate the influence of acute static stretching on the ankle joint position sense of soccer players.

DETAILED DESCRIPTION:
This crossover randomized controlled trial will include semi-professional soccer players. All participants will perform 3 conditions: two experimental conditions, of static stretching of the gastrocnemius and tibialis anterior muscles, for 30 seconds or 90 seconds; and a control condition (rest). Ankle joint position sense of the dominant limb will be assessed before and immediately after the conditions for the range of 20º of plantar flexion by active repositioning, and using a video camera. Absolute, relative and variable angular errors will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* male soccer players from the senior level
* aged between 18 and 30 years old
* with normal plantar flexion range of motion
* without history of lower limb injuries in the last 6 months

Exclusion Criteria:

* those with cardiorespiratory, vestibular or neurological diseases
* with bone or joint deformities in the lower limb
* cerebral concussion in the last 3 months
* history of lower limb surgery
* those with positive ankle integrity tests (anterior drawer test, talus tilt test and external rotation stress test)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Absolute angular error | Change from Baseline (Before) to Immediately after interventions or control (After)
  The absolute value of the difference between the target range and the achieved range
Relative angular error | Change from Baseline (Before) to Immediately after interventions or control (After)
  The arithmetic difference between the target range and the range achieved
Variable angular error | Change from Baseline (Before) to Immediately after interventions or control (After)
  The standard deviation of the 3 repositionings

CONTACTS AND LOCATIONS:
Overall Officials: Joana Azevedo, PhD, Principal Investigator — Escola Superior de Saúde Fernando Pessoa
Locations (1):
- Escola Superior de Saúde Fernando Pessoa, Porto, Portugal

REFERENCES:
- [Derived] Azevedo J, Moreira A, Moreira-Silva I, Cardoso R, Seixas A. The influence of acute static stretching on the ankle joint-position sense of soccer players: A randomized controlled crossover trial. J Bodyw Mov Ther. 2025 Jun;42:1011-1016. doi: 10.1016/j.jbmt.2025.03.022. Epub 2025 Mar 4. PMID 40325629